CLINICAL TRIAL: NCT04384328
Title: Evaluation of an Early Support Programme in Orthophony : the PAPEV-ortho Study
Brief Title: Evaluation of an Early Support Programme in Orthophony
Acronym: PAPEV-ortho
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: rate of inclusions too low
Sponsor: Centre Hospitalier Sud Francilien (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2018-A01898-47
Record Dates: First submitted 2020-02-06; First posted 2020-05-12 (Actual); Last update posted 2023-02-17 (Actual); Status verified 2022-11

CONDITIONS: Language Development Disorders; Preterm Birth
Keywords: language Development; communication Development; preterm infant; orthophony
MeSH Terms: conditions — Language Development Disorders; Premature Birth

STUDY DESIGN:
Intervention Model Description: Prospective, interventionnal with minimal risks and constraints, multicentric, non-randomized, open study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early Support Programme in Orthophony (Experimental): Early support in speech therapy lasts between 6 months and 24 months of corrected age. It includes 10 to 20 sessions depending on the child's needs. These sessions are conducted by a speech-language pathologist from the RPSOF-ASNR network, trained in the issues specific to the very premature child and the network's tools.
  Interventions: Other: Early Support Programme in Orthophony
- Standard Care (No Intervention): Standard follow-up within the RPSOF-ASNR network, without systematic speech therapy sessions.

INTERVENTIONS:
Other: Early Support Programme in Orthophony — Early support in speech therapy lasts between 6 months and 24 months of corrected age. It includes 10 to 20 sessions depending on the child's needs. These sessions are conducted by a speech-language pathologist from the RPSOF-ASNR network, trained in the issues specific to the very premature child and the network's tools.
  Arms: Early Support Programme in Orthophony

SUMMARY:
Prospective, interventionnal with minimal risks and constraints, multicentric, non-randomized, open study, to measure the impact of an early support programme in speech and language therapy for vulnerable children (PAPEV-ortho), in children born very prematurely or very hypotrophically, on the incidence of language and communication deficits at the corrected age of 2 years.

DETAILED DESCRIPTION:
Prospective, interventionnal with minimal risks and constraints, multicentric, non-randomized, open study, to measure the impact of an early support programme in speech and language therapy for vulnerable children (PAPEV-ortho), in children born very prematurely or very hypotrophically, on the incidence of language and communication deficits at the corrected age of 2 years.

Parents of eligible children are informed of the study either during the hospitalization of the neonatal newborn by a hospital physician, or during a consultation performed during the first 6 months by a pilot physician from the RPSOF-ASNR network, hospital or private practitioner. Parents who agree that the data collected about their child may be used in the study sign a written declaration of free and informed consent.

The Early Support Programme in orthophony (PAPEV-ortho) is systematically proposed to families with possible access to a language therapist in the network.

Early support in speech therapy lasts between 6 months and 24 months of corrected age. It includes 10 to 20 sessions depending on the child's needs. These sessions are conducted by a speech-language pathologist from the RPSOF-ASNR network, trained in the issues specific to the very premature child and the network's tools. The support focuses on:

* the development of parental sensitivity and receptivity
* the development of parental reactivity
* optimization of communication sequences in routine acts and play
* the development of the child's intentionality in play and routine acts
* support for verbal and non-verbal oral communication The participation of the child and his or her parents in the study ends at the end of the consultations and evaluations carried out at 24 months of corrected age.

Children within the group that followed the PAPEV-ortho program will be compared to children who did not benefit from this program.

ELIGIBILITY:
Inclusion Criteria:

* Premature birth < 32 weeks of amenorrhea
* or premature birth with intrauterine growth restriction (IUGR) < P3
* corrected age ≤ 6 months at the time of inclusion
* affiliation to a social security system + mutual insurance

Exclusion Criteria:

* genetic pathology
* ongoing developmental care: psychomotricity or speech therapy
* neuromuscular pathology affecting oral and facial motor skills
* severe oral disorders: feeding by gastric tube or gastrostomy
* severe sensory, auditory or visual impairment
* neither of the 2 French-speaking parents

Max Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 76 (Actual)
Dates: Start 2019-11-27 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Score in the Ages & Stages Questionnaires communication domain at 24 months of corrected age. | at 24 months of corrected age
  Percentage of children with a score of ≤ 45 in the communication domain of the Ages & Stages Questionnaires questionnaire (from 0=worst to 60=best) at 24 months of corrected age

SECONDARY OUTCOMES:
Failure rate of implementation of the early support program in speech-language pathology or early drop-out. | at 24 months of corrected age
  Early drop-out is defined by 3 or less sessions.
Score in the Ages & Stages Questionnaires communication domain at 12 and 18 months of corrected age. | at 12 and 18 months of corrected age.
  The Ages & Stages Questionnaires is a parental questionnaire that is strongly correlated with traditional developmental tests. The Ages & Stages Questionnaires communication domain takes into account receptive and expressive language, includes 6 questions, and ranges from 0 (worst) to 60 (best).
score at Inventaire Français du Développement Communicatif questionnaire at 12, 18 and 24 months of corrected age | at 12, 18 and 24 months of corrected age
  The IFDC questionnaire is a recommended tool for monitoring and early detection of language deficits. It is expressed as a percentile (0=worst, 100=best).
Score at Communication and Symbolic Behavior Scales questionnaire at 12 and 24 months of corrected age | at 12 and 24 months of corrected age
  The Communication and Symbolic Behavior Scales qestionnaire is a tool for screening for communication disorders and interactions. It ranges from 0 (worst) tro 57 (best).

CONTACTS AND LOCATIONS:
Overall Officials: Michèle Granier, MD, Study Director — Centre Hospitalier Sud Francilien; Véronique Zupan-Simunek, MD, Principal Investigator — Hôpital Antoine Béclère
Locations (4):
- France (4):
  - Hôpital Antoine Béclère, Clamart
  - Centre Hospitalier Louis Mourier, Colombes
  - Centre Hospitalier Sud Francilien, Corbeil-Essonnes
  - Centre Hospitalier Rives de Seine, Neuilly-sur-Seine

REFERENCES:
- [Result] Pierrat V, Marchand-Martin L, Arnaud C, Kaminski M, Resche-Rigon M, Lebeaux C, Bodeau-Livinec F, Morgan AS, Goffinet F, Marret S, Ancel PY; EPIPAGE-2 writing group. Neurodevelopmental outcome at 2 years for preterm children born at 22 to 34 weeks' gestation in France in 2011: EPIPAGE-2 cohort study. BMJ. 2017 Aug 16;358:j3448. doi: 10.1136/bmj.j3448. PMID 28814566
- [Result] Nishimura T, Takei N, Tsuchiya KJ, Asano R, Mori N. Identification of neurodevelopmental trajectories in infancy and of risk factors affecting deviant development: a longitudinal birth cohort study. Int J Epidemiol. 2016 Apr;45(2):543-53. doi: 10.1093/ije/dyv363. Epub 2016 Feb 13. PMID 26874928
- [Result] Sansavini A, Guarini A, Savini S, Broccoli S, Justice L, Alessandroni R, Faldella G. Longitudinal trajectories of gestural and linguistic abilities in very preterm infants in the second year of life. Neuropsychologia. 2011 Nov;49(13):3677-88. doi: 10.1016/j.neuropsychologia.2011.09.023. Epub 2011 Sep 21. PMID 21958647
- [Result] van Noort-van der Spek IL, Franken MC, Weisglas-Kuperus N. Language functions in preterm-born children: a systematic review and meta-analysis. Pediatrics. 2012 Apr;129(4):745-54. doi: 10.1542/peds.2011-1728. Epub 2012 Mar 19. PMID 22430458
- [Result] Marchman VA, Fernald A. Speed of word recognition and vocabulary knowledge in infancy predict cognitive and language outcomes in later childhood. Dev Sci. 2008 May;11(3):F9-16. doi: 10.1111/j.1467-7687.2008.00671.x. PMID 18466367
- [Result] Stolt S, Lind A, Matomaki J, Haataja L, Lapinleimu H, Lehtonen L. Do the early development of gestures and receptive and expressive language predict language skills at 5;0 in prematurely born very-low-birth-weight children? J Commun Disord. 2016 May-Jun;61:16-28. doi: 10.1016/j.jcomdis.2016.03.002. Epub 2016 Mar 9. PMID 26999726
- [Result] Marchman VA, Loi EC, Adams KA, Ashland M, Fernald A, Feldman HM. Speed of Language Comprehension at 18 Months Old Predicts School-Relevant Outcomes at 54 Months Old in Children Born Preterm. J Dev Behav Pediatr. 2018 Apr;39(3):246-253. doi: 10.1097/DBP.0000000000000541. PMID 29309294
- [Result] Boyer J, Flamant C, Boussicault G, Berlie I, Gascoin G, Branger B, N'Guyen The Tich S, Roze JC. Characterizing early detection of language difficulties in children born preterm. Early Hum Dev. 2014 Jun;90(6):281-6. doi: 10.1016/j.earlhumdev.2014.03.005. Epub 2014 Apr 13. PMID 24726534
- [Result] Sanchez K, Spittle AJ, Slattery JM, Morgan AT. Oromotor Feeding in Children Born Before 30 Weeks' Gestation and Term-Born Peers at 12 Months' Corrected Age. J Pediatr. 2016 Nov;178:113-118.e1. doi: 10.1016/j.jpeds.2016.07.044. Epub 2016 Sep 5. PMID 27609073
- [Result] Telford EJ, Fletcher-Watson S, Gillespie-Smith K, Pataky R, Sparrow S, Murray IC, O'Hare A, Boardman JP. Preterm birth is associated with atypical social orienting in infancy detected using eye tracking. J Child Psychol Psychiatry. 2016 Jul;57(7):861-8. doi: 10.1111/jcpp.12546. Epub 2016 Mar 2. PMID 26934180
- [Result] Eeles AL, Anderson PJ, Brown NC, Lee KJ, Boyd RN, Spittle AJ, Doyle LW. Sensory profiles obtained from parental reports correlate with independent assessments of development in very preterm children at 2 years of age. Early Hum Dev. 2013 Dec;89(12):1075-80. doi: 10.1016/j.earlhumdev.2013.07.027. Epub 2013 Aug 24. PMID 23978398
- [Result] Zuccarini M, Guarini A, Savini S, Iverson JM, Aureli T, Alessandroni R, Faldella G, Sansavini A. Object exploration in extremely preterm infants between 6 and 9 months and relation to cognitive and language development at 24 months. Res Dev Disabil. 2017 Sep;68:140-152. doi: 10.1016/j.ridd.2017.06.002. Epub 2017 Aug 3. PMID 28779627
- [Result] Charkaluk ML, Truffert P, Fily A, Ancel PY, Pierrat V; Epipage study group. Neurodevelopment of children born very preterm and free of severe disabilities: the Nord-Pas de Calais Epipage cohort study. Acta Paediatr. 2010 May;99(5):684-9. doi: 10.1111/j.1651-2227.2010.01695.x. PMID 20491713
- [Result] Crunelle D, Le Normand MT, Delfosse MJ. [Oral and written language production in prematures children: results in 7 1/2-year-old]. Folia Phoniatr Logop. 2003 May-Jun;55(3):115-27. doi: 10.1159/000070723. French. PMID 12771463
- [Result] Forcada-Guex M, Pierrehumbert B, Borghini A, Moessinger A, Muller-Nix C. Early dyadic patterns of mother-infant interactions and outcomes of prematurity at 18 months. Pediatrics. 2006 Jul;118(1):e107-14. doi: 10.1542/peds.2005-1145. PMID 16818525
- [Result] Spittle A, Orton J, Anderson PJ, Boyd R, Doyle LW. Early developmental intervention programmes provided post hospital discharge to prevent motor and cognitive impairment in preterm infants. Cochrane Database Syst Rev. 2015 Nov 24;2015(11):CD005495. doi: 10.1002/14651858.CD005495.pub4. PMID 26597166